CLINICAL TRIAL: NCT06328660
Title: Refitting Biofinity Multifocal Contact Lens Wearer With MyDay Multifocal Contact Lenses
Brief Title: Refitting Multifocal Contact Lens Wearers With a Different Multifocal Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision International Limited (CVIL) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EX-MKTG-155
Record Dates: First submitted 2024-03-12; First posted 2024-03-25 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-07

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens 1 (Experimental): All participants wore Lens 1 for 14 ± 3 days (Period 1)
  Interventions: Device: Lens 1
- Lens 2 (Experimental): All participants wore Lens 2 for 14 ± 3 days (Period 2)
  Interventions: Device: Lens 2

INTERVENTIONS:
Device: Lens 1 — Frequent replacement silicone hydrogel contact lens for 14 ± 3 days on a daily disposable wearing modality
  Arms: Lens 1
Device: Lens 2 — Daily disposable silicone hydrogel contact lens for 14 ± 3 days on a daily disposable wearing modality
  Arms: Lens 2

SUMMARY:
The purpose of this study was to compare ease of handling and vision acuity of two multifocal contact lenses to correct presbyopia that are currently CE marked and on the UK market.

DETAILED DESCRIPTION:
This was an interventional, prospective, open label, sequential design study. Participants wore each study contact lens on a daily disposable wearing modality for 14 ± 3 days and attended the clinic for a total of three study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 years and older;
2. Current multifocal contact lens wearer (other than MyDay® multifocal but can include Biofinity® multifocal);
3. Spectacle refraction:

   * Distance: Sphere: -6.00D to + 4.00D
   * Astigmatism: 0.00D to -0.75D
   * Near Addition: Low +0.75D to +1.25D; Medium +1.50D and +1.75D; High +2.00D to +2.50D
4. Best corrected visual acuity of at least 20/25 in each eye. - The prospective participants will be given a Participant Information Sheet to read and an Informed Consent Form to sign prior to any evaluation.

Exclusion Criteria:

To be eligible as a participant, each candidate shall be free of any ocular or medical condition that may affect the results of this study. The following are specific criteria that exclude a candidate from enrolment in this study:

1. Acute and subacute inflammation or infection of the anterior chamber of the eye.
2. Any eye disease, injury or abnormality that affects the cornea, conjunctiva or eyelids that would contraindicate contact lens wear;
3. Corneal hypoesthesia (reduced corneal sensitivity), if not aphakic
4. Severe insufficiency of lacrimal secretion (dry eyes).
5. Any systemic disease that may affect the eye or may be exaggerated by wearing contact lenses (e.g. acne and eczema).
6. Allergic reactions of ocular surfaces or adnexa that may be induced or exaggerated by wearing contact lenses or use of contact lens solutions
7. Any active corneal infection (bacterial, fungal, protozoal or viral).
8. Newly prescribed (within the past 30 days) use of some systemic medications (such as antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers, stimulants, anti-depressants, anti-psychotics, oral contraceptives) or new prescription eyedrops which is not rewetting/lubricating eyedrops for which contact lens wear could be contraindicated as determined by the investigator;
9. Monocular participants (only one eye with functional vision) or participants fit with only one contact lens;
10. Subjects with slit lamp findings greater than grade 1 (e.g. edema, infiltrates, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival, anterior segment inflammation) as per ISO 11980, any previous history or signs of a contact lens related corneal inflammatory event (past corneal ulcers), or any other ocular abnormality that may contraindicate contact lens wear at the enrolment visit;
11. History of corneal refractive surgery
12. Enrolment of the family members of the investigator, family members of the investigator's staff, or individuals living in the households of these individuals.
13. Current wearer of the test contact lens, MyDay® Multifocal.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Guillon, PhD FCOptom, Principal Investigator — mguillon@otg.co.uk
Locations (1):
- Ocular Technology Group - International, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 67 potential participants were screened, one participant did not fulfil the entry criteria (prescription out of range).
Groups:
- Frequent Replacement Silicone Hydrogel Contact Lens (Lens 1): All participants wore Lens 1 for 14 ± 3 days (Period 1)
- Daily Disposable Silicone Hydrogel Contact Lens (Lens 2): All participants wore Lens 2 for 14 ± 3 days (Period 2)
Period: Lens 1, 14 ± 3 Days
Arm/Group | Frequent Replacement Silicone Hydrogel Contact Lens (Lens 1) | Daily Disposable Silicone Hydrogel Contact Lens (Lens 2)
Started | 66 | 0 (All participants received Lens 1 in Period 1.)
Completed | 66 | 0
Not Completed | 0 | 0
Period: Lens 2, 14 ± 3 Days
Arm/Group | Frequent Replacement Silicone Hydrogel Contact Lens (Lens 1) | Daily Disposable Silicone Hydrogel Contact Lens (Lens 2)
Started | 0 (All participants received Lens 2 in Period 2.) | 66
Completed | 0 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes study participants that completed all study visits
Arm/Group | All Study Participants
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Lens Handling
Description: The ease of contact lens insertion and removal over the week preceding the follow-up visit measured on a 100-point visual analog scale, where 0=Very difficult, Painful and 100=Very easy, Can't feel the lenses
Time Frame: 1 week
Measure: Median (Standard Deviation); unit: score on a scale
Groups:
- Lens 1: Participants that received Lens 1
- Lens 2: Participants that received Lens 2
Arm/Group | Lens 1 | Lens 2
Number analyzed (Participants) | 66 | 66
score on a scale | 96.0 (15.5) | 90.0 (21.0)

2. Secondary Outcome: Overall logMAR Visual Acuity - Dominant Eye
Description: The mean logMAR visual acuity of the dominant eye calculated as the mean of distance, intermediate, and near logMAR visual acuities. This value was recorded at the follow-up visit.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Lens 1 | Lens 2
Number analyzed (Participants) | 66 | 66
logMAR | 0.01 (0.09) | 0.01 (0.09)

3. Secondary Outcome: Overall logMAR Visual Acuity - Non-Dominant Eye
Description: The mean logMAR visual acuity of the non-dominant eye calculated as the mean of distance, intermediate, and near logMAR visual acuities. This value was recorded at the follow-up visit.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Lens 1 | Lens 2
Number analyzed (Participants) | 66 | 66
logMAR | 0.01 (0.07) | 0.00 (0.08)

4. Secondary Outcome: Overall logMAR Visual Acuity - Binocular
Description: The mean binocular logMAR visual acuity calculated as the mean of distance, intermediate, and near logMAR visual acuities. This value was recorded at the follow-up visit.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Lens 1 | Lens 2
Number analyzed (Participants) | 66 | 66
logMAR | -0.05 (0.07) | -0.05 (0.07)

ADVERSE EVENTS:
Time Frame: Duration of the study, approximately 1 month
Arm/Group | Lens 1 | Lens 2
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 4/66 | 6/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lens 1 (N=66) | Lens 2 (N=66)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Flu (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Itchy Eye (Eye disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Common Cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT06328660/Prot_SAP_000.pdf